CLINICAL TRIAL: NCT07039864
Title: A Novel Strategy for Evaluating Gallbladder Contraction Function by Ultrasound: A Prospective, Single-Center, Single-Blind, Cross-Over Trial
Brief Title: A Novel Strategy for Evaluating Gallbladder Contraction Function by Ultrasound
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Responsible Party: Principal Investigator, Wenbo Meng, Director of Surgery, Hepatopancreatobiliary Surgery Institute of Gansu Province
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Gallbladder Function
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Gallbladder; Functional Disturbance
Keywords: Gallbladder; Function; Ultrasound; Fatty Acids

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Accept A processing first, then accept B processing, One week interval (Experimental): A processing: Fasting gallbladder ultrasound in the morning and measure the size of the gallbladder. Immediately take one protein bar orally, and then take 50 milliliters of functional fatty acids orally. Review the gallbladder ultrasound and measure the size of the gallbladder at 1 hour and 1.5 hours.
  Interventions: Diagnostic Test: protein bar first
- Accept B processing first, then accept A processing, One week interval (Active Comparator): B processing: Fasting gallbladder ultrasound in the morning and measure the size of the gallbladder. Immediately ingest two fried eggs orally. Review the gallbladder ultrasound and measure the size of the gallbladder at 1 hour and 1.5 hours.
  Interventions: Diagnostic Test: fried eggs first

INTERVENTIONS:
Diagnostic Test: protein bar first — Take protein bar(after one week fried eggs intake) to evaluate the size of the gallbladder with ultrasound
  Arms: Accept A processing first, then accept B processing, One week interval
Diagnostic Test: fried eggs first — Take fried eggs (after one week protein bar intake) to evaluate the size of the gallbladder with ultrasound
  Arms: Accept B processing first, then accept A processing, One week interval

SUMMARY:
This study is a prospective, single-center, single-blind, cross-over trial conducted at a tertiary hospital, aiming to determine the evaluation of oral functional fatty acids on gallbladder contractile function.

DETAILED DESCRIPTION:
The most commonly used methods for assessing gallbladder emptying function are radionuclide imaging and ultrasonography. Radionuclide imaging, although effective, has several limitations including lengthy examination time, relatively high costs, and reliance on radioactive isotopes, which has led to its gradual replacement by ultrasonography in clinical practice. Ultrasonography offers significant advantages as a non-invasive modality, providing highly accurate functional evaluations through quantitative analysis. This method objectively reflects gallbladder contraction and emptying capabilities with minimal human interference and demonstrates high reproducibility. Assessment of gallbladder contractile function requires the patient to perform an ultrasound examination on an empty stomach to measure the length, transverse and anterior and posterior diameters of the gallbladder, thus calculating the volume of the fasting gallbladder. The patient is then given a fat meal (usually 2 fried eggs), and the ultrasound examination is performed again 60 minutes after eating to measure the volume of the gallbladder. Gallbladder contractile function is assessed by comparing changes in gallbladder volume on an empty stomach and after a meal. Under normal circumstances, the contraction rate of the gallbladder should reach a certain level. It is generally considered normal to have a contraction rate greater than 30% -50%. However, eating a fat meal, because the fat content of the food itself cannot be accurately determined, will bring inaccurate factors to the evaluation of gallbladder contractile function, such as eating fried eggs, because the variety, size, and quantity of eggs are different, the cooking oil used is different, and the amount of cooking oil remaining on the fried eggs is also different resulting in a large difference in the content of fat in the human body when orally ingested, ultimately leading to an inaccurate evaluation of gallbladder contractile function. Notably, cholesterol in fried eggs may intensify clinical manifestations of cholecystitis, thus necessitating caution when recommending fried eggs to patients with active gallbladder inflammation. Therefore, a prospective, single-center, single-blind, cross-over trial was conducted to verify whether oral functional fatty acids can be used to effectively evaluate gallbladder contractile function.

ELIGIBILITY:
Inclusion Criteria:

* Ultrasound assessment identifies people with normal biliary tract structure

Exclusion Criteria:

* History of Endoscopic Retrograde Cholangiopancreatography
* Previous gallstone removal surgery with gallbladder preservation
* History of acute or chronic pancreatitis, cholangitis
* Mirizzi Syndrome
* History of gastrointestinal surgery
* Gastrointestinal obstruction
* Dysfunction of the sphincter of Oddi
* Gallbladder neck polyps
* Abnormal gallbladder structure
* Gallbladder mass
* Biliary infection or stones
* Congenital biliary abnormalities
* Biliary injury or surgery
* Biliary tumors
* Gastrointestinal bleeding, liver cirrhosis, or other malignant diseases
* Significant arrhythmia, bradycardia, or atrioventricular block
* Severe hypertension, liver or kidney insufficiency
* Immune, endocrine, hematological, or mental disorders
* Severe cerebrovascular disease
* Allergy to relevant foods
* Pregnant or breastfeeding women
* Unwillingness or inability to consent to participation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2025-06-26 (Actual); Primary Completion 2025-12-20 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
Gallbladder Volume | 1 day
  Ultrasound will be used to measure the volume of the gallbladder on the empty stomach and after the intervention. Formula for Ultrasound Measurement of Gallbladder Volume (L × W × D × 0.52)
Gallbladder contraction rate | 1 day
  The volume of the gallbladder on an empty stomach minus the volume of the gallbladder after the intervention, divided by the volume of the gallbladder on an empty stomach, and finally multiplied by 100%（A-B/A%） Gallbladder contraction rate after 1 hour of oral administration of functional fatty acids with Complete gallbladder emptying100% or Good gallbladder contractility50% or Abnormal gallbladder contractility0%

SECONDARY OUTCOMES:
Presence of Abdominal Pain Post-Intervention | 7 days
  If abdominal pain is present, it will be assessed using the Numerical Rating Scale (NRS) within 0-10, The higher the score, the more serious it is
Occurrence of Acute Pancreatitis Post-Intervention | 7 days
  Pain and Amy 3 times as normal
Occurrence of Gastrointestinal Bleeding Post-Intervention | 7 days
  Black stool or decrease of hemoglobin
Nausea, Vomiting, and Diarrhea Post-Intervention | 7days
  Frequency of Nausea, Vomiting, and Diarrhea Post-Intervention

CONTACTS AND LOCATIONS:
Overall Officials: Wenbo Meng, M.D. Ph. D., Principal Investigator — Hepatopancreatobiliary Surgery Institute of Gansu Province
Locations (1):
- Hepatopancreatobiliary Surgery Institute of Gansu Province, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ai XN, Wang TF, Zhang Q, Ouyang CG, Wu ZY. Changes in Gallbladder Contractile Function and its Influencing Factors After Minimally Invasive Gallbladder-Preserving Surgery for Cholecystitis With Incarcerated Gallstones. Front Surg. 2022 Jul 14;9:926141. doi: 10.3389/fsurg.2022.926141. eCollection 2022. PMID 35910468
- [Result] Deinega VG, Medvedev VV, Polishchuk LM. [The evaluation of gallbladder contractile function and the ultrasonic signs of chronic noncalculous cholecystitis]. Lik Sprava. 1992 Jun;(6):103-6. Russian. PMID 1455813